CLINICAL TRIAL: NCT05580588
Title: A Phase 2 Multicenter, Open-Label Study of the CDK4/6 Inhibitor SPH4336 in Subjects With Locally Advanced or Metastatic Liposarcomas
Brief Title: Open-Label Study of the CDK4/6 Inhibitor SPH4336 in Subjects With Locally Advanced or Metastatic Liposarcomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Although no safety issues with SPH4336 were identified, efficacy in liposarcoma patient was less than anticipated.
Sponsor: Shanghai Pharma Biotherapeutics USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH4336-US-01
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Liposarcoma, Dedifferentiated
Keywords: CDK4/6 inhibitor
MeSH Terms: conditions — Liposarcoma

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPH4336 (Experimental): 400 mg (2 - 200 mg tablets) PO QD
  Interventions: Drug: SPH4336

INTERVENTIONS:
Drug: SPH4336 — 400 mg SPH4336 PO QD

SUMMARY:
Study SPH4336-US-01 is an open-label (no placebo), multicenter clinical trial to evaluate the safety, blood levels (pharmacokinetics) and preliminary anti-tumor effects of SPH4336, a selective enzyme blocker, in patients with specific types of liposarcomas (tumors expressing the target of the study drug).

DETAILED DESCRIPTION:
Study SPH4336-US-01 is a multicenter, non-randomized, open-label Phase 2 study of SPH4336 with a safety lead-in in subjects with CDK4-positive liposarcomas (dedifferentiated or well-differentiated/dedifferentiated liposarcomas). SPH4336 is an orally administered, molecularly targeted chemotherapy drug called a cyclin-dependent kinase inhibitor (CDK4/6 inhibitor), which acts to block the ability of cancer cells to divide and thus prevents tumors from growing. SPH4336 (tablets) will be administered orally once each day in successive 28-day cycles until demonstration of progressive disease or the development of unacceptable toxicity.

The study will incorporate a safety lead-in for the initial 10 subjects. Safety will be evaluated after 10 subjects (minimum 1 cycle completed) by a Safety Review Committee (SRC). The study will be stopped if unacceptable toxicity is observed in more than 2 subjects.

Tumor assessments according to RECIST v1.1 will be performed at baseline and every 6 weeks (from Cycle 1, Day 1 (C1D1)) for 36 weeks, then every 12 weeks thereafter. Plasma samples for pharmacokinetics will be collected in all subjects. Baseline (pretreatment) tumor tissue (archival or fresh) will be collected from all subjects to confirm histologically a liposarcoma with a dedifferentiated component and CDK4 positivity. Tumor tissue biomarkers (e.g., phospho-Rb, Ki-67) will be analyzed in the first 10 study subjects in baseline (pretreatment) and C1D15 tumor tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* ≥ 18 years of age
* ECOG performance status 0 or 1
* Histologically confirmed, locally advanced or metastatic sarcoma

  * Dedifferentiated or well-differentiated/dedifferentiated liposarcomas
* No more than 3 prior lines of treatment
* Evidence of progression as evidenced by at least one of the following within the past 3 months:

  * An increase of at least 20% in measurable tumors
  * The appearance of new lesions
  * Unequivocal progression of non-measurable lesions
* Measurable disease per RECIST v1.1
* If residual treatment-related toxicity from prior therapy:

  * All treatment-related toxicity resolved to Grade 1 or baseline (alopecia excepted)
* ANC ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Hgb ≥ 9.0 g/dL (in the absence of pRBC transfusion over the prior 4 weeks)
* Estimated glomerular filtration rate of ≥ 60 mL/min (based on the Cockcroft and Gault formula for individualized estimates of GFR)
* Total bilirubin ≤ 1.5 x the Upper Limit of Normal (ULN) or ≤ 3 x ULN if known Gilbert's disease
* AST and ALT ≤ 3 x ULN or ≤ 5 x ULN if malignant involvement of the liver
* Sterile or willing to use effective contraception (approved hormonal contraceptive such as oral contraceptives, patches, implants, injections, rings or hormonally-impregnated intrauterine device (IUD), or an IUD in women of childbearing potential and a condom in men) during the study and for 3 months following the last dose of study drug
* Availability of archived tumor tissue or willingness to undergo a baseline tumor biopsy, and in the first 10 study subjects, to determine baseline tumor biomarker levels and a willingness to undergo a second tumor biopsy at C1D15 to assess treatment-induced changes in tumor biomarker levels

Exclusion Criteria:

* Prior treatment with a CDK4/6-targeted agent
* Patient's tumor known to be CDK4 negative
* Anticancer therapy (e.g., chemotherapy, biologics, irradiation) within 14 days or 5 half-lives (whichever is greater) of screening
* Major surgery within 28 days of screening
* Requirement for systemic treatment with strong CYP3A4 inhibitors or inducers of CYP3A4 at study entry
* Central nervous system metastases or leptomeningeal disease, unless appropriately treated and neurologically stable without steroids for ≥ 28 days
* Other malignancy unless disease-free for ≥ 2 years and not expected to relapse or require treatment during study participation
* Active systemic infection or severe localized infection
* Known HIV-positive with CD4+ cell counts < 350 cells/uL or a history of an AIDS-defining opportunistic infection
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with viral load above the limit of quantification
* Active COVID-19 infection
* Major cardiac abnormalities (e.g., uncontrolled angina, unstable arrhythmias, myocardial infarction, NYHA Class ≥ 3 CHF) ≤ 6 months of C1D1
* Persistent (3 ECGs ≥ 5 mins apart) prolongation of the QTcF (Fridericia) > 470 msec
* [Females] Pregnant or nursing
* Any other medical or psychiatric condition, or laboratory abnormality that would result in an unacceptable risk with study participation
* Presence of active gastrointestinal disease or other condition expected to interfere significantly with absorption, distribution, metabolism or excretion of oral therapy (e.g., ulcerative disease, uncontrolled nausea, vomiting, chronic diarrhea, malabsorption syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Locke, PhD, Study Director — Shanghai Pharma Biotherapeutics USA Inc.
Locations (9):
- United States (9):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Seidman Cancer Center, University Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated for efficacy lower than company standards
Pre-assignment Details: Study participants required to meet all I/E criteria prior to enrollment
Period: Overall Study
Arm/Group | SPH4336
Started | 14
Completed | 2
Not Completed | 12
Not completed — Lack of Efficacy | 12

BASELINE CHARACTERISTICS:
Arm/Group | SPH4336
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 12 Weeks
Description: Number of total patients who are progression-free, as defined as RECIST v1.1 (a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions), at 12 weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SPH4336
Number analyzed (Participants) | 14
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for individual patients from signing of the Informed Consent until their discontinuation from the study due to disease progression, pregnancy, serious adverse events, death, or termination of the study by the Sponsor (on average, less than 1 year).
Arm/Group | SPH4336
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPH4336 (N=14)
elevated ALT (Investigations) | 2 (2)
elevated AST (Investigations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPH4336 (N=14)
diarrhea (Gastrointestinal disorders) | 10 (10) — Gr 1
vomiting (Gastrointestinal disorders) | 2 (2) — Gr 1
blood creatinine (Investigations) | 2 (2) — Gr 1
neutrophil count decreased (Investigations) | 2 (2) — Gr 3
fatigue (General disorders) | 5 (5) — Gr 1
decreased appetite (General disorders) | 2 (2) — Gr 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT05580588/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05580588/SAP_001.pdf